CLINICAL TRIAL: NCT02159209
Title: The Genetic Contribution to Drug Induced Renal Injury: The Drug Induced Renal Injury Consortium (DIRECT)
Brief Title: The Drug Induced Renal Injury Consortium
Acronym: DIRECT
Status: Completed | Type: Observational
Sponsor: Ravindra Mehta (Other)
Collaborators: International Serious Adverse Event Consortium (Unknown)
Responsible Party: Sponsor-Investigator, Ravindra Mehta, Professor of Clinical Medicine, University of California, San Diego
Organization: University of California, San Diego (Other)
Other Study IDs: 121651
Record Dates: First submitted 2013-09-26; First posted 2014-06-09 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-04

CONDITIONS: Acute Kidney Injury; Adverse Drug Reaction; Acute Kidney Failure; Kidney Failure; Kidney Disease
Keywords: Acute Kidney Injury; Adverse Drug Reaction; Acute Kidney Failure; Kidney; Kidneys
MeSH Terms: conditions — Acute Kidney Injury; Drug-Related Side Effects and Adverse Reactions; Renal Insufficiency; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Plasma, serum, and urine stored for further analysis of biomarkers
  * Urinary chemistry
  * Urinary microscopy
  * DNA sample
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Drug Induced Renal Injury (DIRI): This is a prospective observational cohort study of patients who have developed acute kidney injury Stage 2 or a glomerular disorder following exposure to specific drugs that have been associated with DIRI.

SUMMARY:
Some medications are known to cause kidney damage because the person is allergic to the medication while others cause direct damage to the kidney because they are toxic at certain concentrations. Risk factors for developing kidney damage have been identified for some medications but not for all. Patients who are exposed to these important medications and develop problems with their kidneys may have some genetic risk. The purpose of this study is to determine the genetic risk factors for drug induced kidney injury. A better understanding of the role of genetics for the development of kidney injury from medications will allow us to better select medications, improve effectiveness of treatment and minimize harm.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 2 years and older
* Exposure to a candidate drug for at least 24 hours (see above)
* Patients who have developed DIRI as defined by the primary criteria
* Written informed consent or assent and consent obtained
* If patient lacks capacity to consent then surrogate consent will be obtained

Exclusion Criteria:

* Patients with a history of or have a kidney transplant
* Patients with a history of or have a bone marrow transplant
* Patients with Chronic Kidney Disease stage 5 (eGFR < 15 mL/min/1.73m2)
* Patients on 3 or more causal drugs
* Patients with no history or time course on drug exposure
* Patient who, in the opinion of the Investigator, is not suitable to participate in the study.
* Unable to obtain written informed consent or assent
* Unable to obtain surrogate consent for patients who lack capacity

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a prospective observational cohort study of patients who have developed DIRI. Patients will be identified through two main approaches;
  1. Recall and review of medical records of patients who were suspected to have DIRI
  2. Concurrent identification of patient under active treatment.
  Patients who developed DIRI in their previous care provided will be identified through a review of kidney biopsy logs or nephrology consults previously made.
Sampling Method: Non-Probability Sample
Enrollment: 634 (Actual)
Dates: Start 2013-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Identify genes that predispose to dose dependent (Type A) or hypersensitivity (Type B) during drug induced nephrotoxicity. | At time of enrollment
  Blood Draw (20 cc) and urine collection (80cc)

SECONDARY OUTCOMES:
To identify specific alterations in drug metabolism pathways that contribute to drug induced renal injury with different drugs. | DNA sample collected at time of enrollment.
  We will perform a GWAS to examine the association of common genetic variants with the development of DIRI. For assessing association between a common SNP and the risk of DIRI, association tests will be undertaken to compare genotype frequencies between cases and controls. We will use logistic regression models under the assumption of an additive genetic model and incorporate potential confounders and covariates. Dominant, recessive models will also be checked through alternative coding of the genotype for SNPs approaching significance.

CONTACTS AND LOCATIONS:
Overall Officials: Ravindra Mehta, MD, Principal Investigator — University of California, San Diego
Locations (18):
- United States (8):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of California, San Diego, San Diego, California
  - Rady Children's Hospital, San Diego, California
  - University of Colorado, Aurora, Colorado
  - University of Michigan, Ann Arbor, Michigan
  - St. Peter's Hospital, Albany, New York
  - Jacobi Medical Center, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
- Universidad del Valle, Cochabamba, Cochabamba, Bolivia
- Hopital Sacre Coeur & Universite de Montreal, Montreal, Quebec, Canada
- Universidad de Los Andes, Santiago, Chile
- India (2):
  - CARE Hospitals, Banjara Hills, Hyderabad
  - Postgraduate Institute of Research, Chandigarh, Chandigarh
- United Kingdom (5):
  - Newcastle University, Newcastle upon Tyne, Tyne and Wear
  - St James's University Hospital, Leeds, West Yorkshire
  - Royal Free Hospital, London
  - Guy's & St Thomas's Hospital, London
  - University of Nottingham, Nottingham

REFERENCES:
- [Background] Mehta RL, Awdishu L, Davenport A, Murray PT, Macedo E, Cerda J, Chakaravarthi R, Holden AL, Goldstein SL. Phenotype standardization for drug-induced kidney disease. Kidney Int. 2015 Aug;88(2):226-34. doi: 10.1038/ki.2015.115. Epub 2015 Apr 8. PMID 25853333
- [Derived] Yousif Z, Awdishu L. Drug-Induced Acute Kidney Injury Risk Prediction Models. Nephron. 2023;147(1):44-47. doi: 10.1159/000526267. Epub 2022 Sep 9. PMID 36088907